CLINICAL TRIAL: NCT01303549
Title: Multicenter, Randomized, Open-label Clinical Trial to Compare Anidulafungin Versus Amphotericin B Safety in High Risk Hepatic Transplant Recipients
Brief Title: Anidulafungin vs Amphotericin B Safety in High Risk Hepatic Transplant Recipients
Acronym: AVALTRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion SEIMC-GESIDA (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GESITRA 0110; 2011-000804-17 (EudraCT Number)
Record Dates: First submitted 2011-02-16; First posted 2011-02-24 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2013-09

CONDITIONS: Liver Disease; Fungal Infection
Keywords: Liver transplantation; Hepatic transplant; Antifungal prophylaxis; Anidulafungin; Liposomal Amphotericin B
MeSH Terms: conditions — Liver Diseases; Mycoses | interventions — Anidulafungin; liposomal amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anidulafungin (Experimental): Anidulafungin IV once a day: initial dose 200 mg/day, following doses 100 mg/day.
  Interventions: Drug: Anidulafungin
- Liposomal Amphotericin B (Active Comparator): Liposomal amphotericin B once a day: 3 mg/kg/day
  Interventions: Drug: Liposomal amphotericin B

INTERVENTIONS:
Drug: Anidulafungin — Anidulafungin once a day for 14 days: initial dose 200 mg/day IV administered in 180 minutes. Following doses 100 mg/day IV administered in 90 minutes.
  Other Names: Ecalta
  Arms: Anidulafungin
Drug: Liposomal amphotericin B — Liposomal amphotericin B once a day for 14 days: 3 mg/kg/day. IV administration during 60 minutes.
  Other Names: AmBisome
  Arms: Liposomal Amphotericin B

SUMMARY:
The study is a randomized, open-label safety study comparing the use of anidulafungin (200 mg i.v. as initial dose and 100 mg/d i.v. in subsequent doses) vs liposomal amphotericin B (3 mg/kg/d i.v.) in hepatic transplant recipients who have high risk of fungal infection.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Signature of ICF
* Negative pregnancy test (women of child bearing potential)
* Patients who comply with at least one of the following (A or B):

A: One of the following criteria (major criteria):

* Re-transplant due to severe dysfunction of a previous hepatic graft
* Requirement of any renal substitutive therapy, including dialysis or hemofiltration
* Fulminant hepatitis requiring hepatic transplant

B: Two of the following criteria (minor criteria):

* Post-transplant renal impairment (defined as CrCl< 50 mL/min) 30 days after transplantation
* Intra surgery blood transfusion of at least 40 units
* Choledochal jejunectomy
* 2 or more Candida sp cultures (nasal, pharynx, rectal) from 48 hours pre- to 48 hours post-hepatic transplant
* Post transplant re-intervention (laparotomy)

Exclusion Criteria:

* Hypersensibility to amphotericin B or candin
* Patients who have received any other antifungal (excluding fluconazole or oral nystatin for a maximum of 7 days)
* Documented or suspected fungal infection
* Pregnant women of women who do not accept to us a valid anticonceptive method
* Any other disease or medical condition that makes the patient not adequate to participate in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Renal impairment/renal function deterioration | 14 days
  Compare the development of renal imparment or deterioration of baseline renal function in hepatic transplat recipients who receive anidulafungin or liposomal amphotericin B
Number of infusion related adverse events | 14 days
  Compare the development of infusion related adverse events in hepatic transplat recipients who receive anidulafungin or liposomal amphotericin B

SECONDARY OUTCOMES:
Treatment discontinuation | 14 days
  Compare the proportion of patiens who discontinue antifungal profilaxis in both arms
Hepatic toxicity | 14 days
  Compare the emergence of hepatic toxicity in both arms
Invasive fungal infection | Week 12 and week 24
  Compare the incidence of early (first 12 weeks) and delayed (until week 24) invasive fungal infection between both arms
Mortality | 24 weeks post transplantation
  Compare the mortality rate (both global and fungal infection related) between both arms 24 weeks after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Cervera, MD, Study Director — Hospital Clinic i Provincial; Asuncion Moreno, MD, Principal Investigator — Hospital Clinic i Provincial; Carmen Fariñas, MD, Principal Investigator — Hospital Marqués de Valdecilla
Locations (12):
- Spain (12):
  - Hospital Reina Sofia, Córdoba, Córdoba
  - Complexo Hospitalario de A Coruña, A Coruña
  - Hospital Clinic i Provincial, Barcelona
  - Hospital de Bellvitge, Barcelona
  - Hospital Vall d'Hebrón, Barcelona
  - Hospital de Cruces, Bilbao
  - Hospital Doce de Octubre, Madrid
  - Hospital Gregorio Marañón, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Carlos Haya, Málaga
  - Hospital Central de Asturias, Oviedo
  - Hospital Marqués de Valdecilla, Santander